CLINICAL TRIAL: NCT04148638
Title: Dr. Pao-Lin Kuo (Department of Obstetrics and Gynecology)
Brief Title: Explore the Role of NLRP7 in the Regulation of Progestereone Induced Decidualization of Human Endometrial Stroma Cells
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: A-ER-102-440
Record Dates: First submitted 2019-10-28; First posted 2019-11-01 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2019-11

CONDITIONS: Inflammatory Response; Abortion, Habitual
MeSH Terms: conditions — Abortion, Habitual

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood

SUMMARY:
The investigators have found that NLRP7 was upregulated and nuclear translocated in an in vitro model of decidualization. Knock-down or overexpression of NLRP7 reduced or enhanced the expression of decidual marker IGFBP-1. NLRP7 was also found to promote progesterone receptor (PR) activity. So, the investigators hypothesized that NLRP7 may regulate progesterone-induced decidualization of human endometrial stromal cells. Part I is to explore how NLRP7 is induced during the decidualization. According to the luciferase activities of NLRP7 promoter luciferase reporter systems, the region from -100 to +37 or from -1200 to -100 had positive or negative regulatory elements, respectively, in the in vitro decidualization. Part II is to explore how NLRP7 contributes the decidualization of endometrial stromal cells. By immunoprecipitations of NLRP7 or PR, the investigators found NLRP7 might involve in the transcriptional complex of PR in the in vitro decidualization. The NLRP7 interacting protein in the co-immunoprecipitations the investigatorsre analyzed by LC/MS-MS. Part III is to explore the effects of NLRP7 mutations on in vitro decidualization and macrophage differentiation.

Comparing to RFP control, the investigators found wild-type NLRP7 enhanced but NLRP7 mutants reduced IGFBP-1 expression in the in vitro decidualization. In the M1 macrophage differentiation of THP-1, wild-type and mutant NLRP7 reduced IL-1β expression compared to the RFP control. Part IV is to explore a role of MPA in macrophage differentiation. MPA drives THP-1 cells a M2-like macrophage differentiation toward a phenotype of decidual macrophages, which promoted in vitro decidualization and trophoblastic invasion, but tolerated TLR ligands stimulations. In conclusion, NLRP7 contributes in vitro decidualization of endometrial stromal cells; NLRP7 mutation may impede in vitro decidualization; NLRP7 may suppress IL-1 expression in M1 macrophage differentiation; MPA drives M2 macrophage differentiation toward a phenotype of decidual macrophage.

DETAILED DESCRIPTION:
The investigators have found that NLRP7 was upregulated and nuclear translocated in an in vitro model of decidualization. Knock-down or overexpression of NLRP7 reduced or enhanced the expression of decidual marker IGFBP-1. NLRP7 was also found to promote progesterone receptor (PR) activity. So, the investigators hypothesized that NLRP7 may regulate progesterone-induced decidualization of human endometrial stromal cells. Part I is to explore how NLRP7 is induced during the decidualization. According to the luciferase activities of NLRP7 promoter luciferase reporter systems, the region from -100 to +37 or from -1200 to -100 had positive or negative regulatory elements, respectively, in the in vitro decidualization. Part II is to explore how NLRP7 contributes the decidualization of endometrial stromal cells. By immunoprecipitations of NLRP7 or PR, the investigators found NLRP7 might involve in the transcriptional complex of PR in the in vitro decidualization. The NLRP7 interacting protein in the co-immunoprecipitations the investigatorsre analyzed by LC/MS-MS. Part III is to explore the effects of NLRP7 mutations on in vitro decidualization and macrophage differentiation. Comparing to RFP control, the investigators found wild-type NLRP7 enhanced but NLRP7 mutants reduced IGFBP-1 expression in the in vitro decidualization. In the M1 macrophage differentiation of THP-1, wild-type and mutant NLRP7 reduced IL-1β expression compared to the RFP control. Part IV is to explore a role of MPA in macrophage differentiation. MPA drives THP-1 cells a M2-like macrophage differentiation toward a phenotype of decidual macrophages, which promoted in vitro decidualization and trophoblastic invasion, but tolerated TLR ligands stimulations. In conclusion, NLRP7 contributes in vitro decidualization of endometrial stromal cells; NLRP7 mutation may impede in vitro decidualization; NLRP7 may suppress IL-1 expression in M1 macrophage differentiation; MPA drives M2 macrophage differentiation toward a phenotype of decidual macrophage.

ELIGIBILITY:
Inclusion Criteria:

Fertility woman 20-50 years-of-age -Hydatidiform Mole or Habitualabortion Exclusion Criteria:NA

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: It is known that NLRP7, a member of the protein family related to innate immunity, is associated with habitual abortion, and it is found that dysfunction of NLRP7 protein may affect endometrial decidualization and facilitate embryo implantation.
Sampling Method: Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
NLRP7 expressed in the decidualized stromal cells of the human endometrium during the first trimester. | 1 day
  The tissue sections of the non-pregnant endometrium (n = 5) or the first trimester endometrium (n = 5) were deparaffinized, rehydrated and stained with NLRP7 antibody. Representative images of NLRP7 immunohistochemistry in the endometrium are shown. The NLRP7 signal was developed with the anti-rabbit HRP antibody and AEC substrate. Staining with the 2nd antibody only served as the negative control. Arrows point to the endometrial stromal cells. NLRP7 dominantly appeared in the swollen decidualized stromal cells of pregnant endometrium, but not in the stromal cells of non-pregnant endometrium (magnification 200X)

CONTACTS AND LOCATIONS:
Overall Officials: Pao-Lin Kuo, MD, Principal Investigator — Department of Obstetrics and Gynecology, National Cheng Kung University Hospital
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan